CLINICAL TRIAL: NCT00430001
Title: A Randomised Phase III Study of Trastuzumab-Docetaxel vs Trastuzumab-Vinorelbine as 1. Line Therapy for Patients With Metastatic HER2 Positive Breast Cancer
Brief Title: Vinorelbine Plus (+) Trastuzumab vs Docetaxel Plus (+) Trastuzumab as 1 Line Treatment for HER2 Positive (+) Metastatic Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish Breast Cancer Cooperative Group (Other)
Collaborators: Hoffmann-La Roche (Industry); Sanofi (Industry)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HERNATA
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Breast Cancer
Keywords: Metastatic breast neoplasm
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Vinorelbine; Trastuzumab

INTERVENTIONS:
Drug: docetaxel
Drug: vinorelbine
Drug: trastuzumab

SUMMARY:
In an open-label randomised phase III-trial patients with metastatic HER2-positive breast cancer naive to chemotherapy with normal organ function and WHO performance status < 3 are randomised to receive either docetaxel 100 mg/m2 i.v. plus trastuzumab 6 mg/kg (8 mg/kg loading dose) q 3 weeks or vinorelbine 30 or 35 mg/m2 days 1+8 plus trastuzumab 6 mg/kg (8 mg/kg loading dose) q 3 weeks. Primary endpoint is time to progression. Secondary endpoints include overall survival, time to treatment failure, response rate, duration of response and toxicity. The study hypothesis is that docetaxel is more efficient than vinorelbine but also more toxic.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic HER2-positive breast cancer
* WHO performance status < 3

Exclusion Criteria:

* Chemotherapy for metastatic breast cancer or adjuvant therapy within 12 months with docetaxel, vinorelbine or trastuzumab
* Severe dyspnoea
* Abnormal organ function including cardiac

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2005-05; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | median

SECONDARY OUTCOMES:
response rate, overall survival, toxicity | Median

CONTACTS AND LOCATIONS:
Overall Officials: Michael Andersson, MD D Med Sci, Principal Investigator — Department of Oncology 5074, Rigshospitalet, 2100 Copenhagen, Denmark
Locations (1):
- Department of Oncology, Rigshospitalet, Copenhagen, Denmark